CLINICAL TRIAL: NCT06581965
Title: The DISTINCT Trial: inDividual, Targeted thrombosIS Prophylaxis Versus the Standard 'One Size Fits All' Approach in Patients Undergoing Total hIp or Total kNee replaCemenT: a National, Multicenter, Randomized, Multi-arm, Open-label Trial.
Brief Title: inDividual, Targeted thrombosIS Prophylaxis Versus the Standard 'One Size Fits All' Approach in Patients Undergoing Total hIp or Total kNee replaCemenT
Acronym: DISTINCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, B.Nemeth, Postdoctoral researcher Clinical epidemiology, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P24.031; 2023-510186-98-00 (EU CTIS Number); U1111-1305-2311 (Registry Identifier: Universal trial number)
Record Dates: First submitted 2024-08-25; First posted 2024-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Venous Thromboembolism; Venous Thromboses; Pulmonary Embolism; Deep Vein Thrombosis
Keywords: Venous thromboembolism; Prophylaxis; Individualized Medicine; Total hip arthroplasty; Total knee arthroplasty; Randomized controlled trial
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: This trial consists of 3 study arms. DISTINCT 1 (low VTE risk <1.0%): randomized (2 arms) DISTINCT 2 (intermediate VTE risk 1.0%-1.5%): observational DISTINCT 3 (high VTE risk >1.5%): randomized (2 arms) Participants will be allocated to a study arm based on their predicted VTE risk which is determined by the TRiP(plasty) score.
Masking Description: Blinded endpoint adjudication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- DISTINCT 1 short duration prophylaxis (Experimental): Patients with a low VTE risk (predicted 3-months postoperative VTE risk <1%) based on the TRiP(plasty) score. (Nemeth, 2024)
  Interventions: Other: Short duration prophylaxis
- DISTINCT 1 control (Active Comparator): Patients with a low VTE risk (predicted 3-months postoperative VTE risk <1%) based on the TRiP(plasty) score. (Nemeth, 2024)
  Interventions: Other: Control
- DISTINCT 2 observational arm (Other): Patients with an intermediate VTE risk (predicted 3-months postoperative VTE risk ≥1%-≤1.5%) based on the TRiP(plasty) score. (Nemeth, 2024)
  Interventions: Other: Control
- DISTINCT 3 extended prophylaxis (Experimental): Patients with a high VTE risk (predicted 3-months postoperative VTE risk >1.5%) based on the TRiP(plasty) score. (Nemeth, 2024)
  Interventions: Other: Higher intensity and longer duration prophylaxis
- DISTINCT 3 control (Active Comparator): Patients with a high VTE risk (predicted 3-months postoperative VTE risk >1.5%) based on the TRiP(plasty) score. (Nemeth, 2024)
  Interventions: Other: Control

INTERVENTIONS:
Other: Short duration prophylaxis — Only during hospitalization: any type of LMWH or DOAC in a prophylactic dose as approved by the Dutch guideline "Antitrombotisch beleid". First dose of LMWH within 6-24h following surgery. First dose of apixaban within 12-24h following surgery. First dose of rivaroxaban 6-10h following surgery. First dose of dabigatran within 1-4h following surgery. The applied type of anticoagulant is according to the local standard use (same type as used for control group).
  Arms: DISTINCT 1 short duration prophylaxis
Other: Higher intensity and longer duration prophylaxis — The use of any thrombocyte aggregation inhibitors should be discontinued 5 days prior to surgery. Day 0-2: any type of LMWH or DOAC in a prophylactic dose as approved by the Dutch guidelines. First dose of LMWH within 6-24h following surgery. First dose of apixaban within 12-24h following surgery. First dose of rivaroxaban 6-10h following surgery. First dose of dabigatran within 1-4h following surgery. The applied type of anticoagulant is according to the local standard use.
  Day 3: Apixaban 5mg b.i.d., continued until 6 weeks after surgery, conditional on the fact that no active bleeding of the surgical wound can be observed. In case of active bleeding, the prophylactic dose of thrombosis prophylaxis is continued. Thereafter, in case no active bleeding has been observed for 24 hours, the 5mg b.i.d. apixaban treatment will be started.
  The 5mg b.i.d. apixaban dose will be adjusted to 2.5mg b.i.d. in case of an impaired kidney function (defined as eGFR 10-30ml/min).
  Arms: DISTINCT 3 extended prophylaxis
Other: Control — 4 weeks: any type of LMWH or DOAC in a prophylactic dose as approved by the Dutch guidelines. First dose of LMWH within 6-24h following surgery. First dose of apixaban within 12-24h following surgery. First dose of rivaroxaban 6-10h following surgery. First dose of dabigatran within 1-4h following surgery. The applied type of anticoagulant is according to the local standard use.
  Other Names: Standard treatment
  Arms: DISTINCT 1 control; DISTINCT 2 observational arm; DISTINCT 3 control

SUMMARY:
After hip or knee replacement all patients receive a standardized treatment with blood thinners, this medication is called thrombosis prophylaxis. However, despite this standard treatment some individuals still develop venous thrombosis (VTE), while others experience bleeding. This indicates that not all patients have the same VTE risk following surgery. Individualizing the amount of thrombosis prophylaxis following surgery might lead to less thrombotic and bleeding events. In this study the investigators individualize the treatment with thrombosis prophylaxis based on the medical history of a patient.

The main questions this study aims to answer are:

Can thrombosis prophylaxis be shortened in patients with a low VTE risk to decrease the risk of bleeding without increasing the risk of VTE? Does an increase in the dose and duration of thrombosis prophylaxis in patients with a high VTE risk reduce the risk of VTE without inducing an unacceptable risk of bleeds?

Researchers will compare both the shortened treatment in low VTE risk patients and the intensified and extended treatment in high VTE risk patients with the standard treatment to assess the risk of VTE and bleeding in comparison to the standard treatment.

Participants will receive 4 questionnaires to evaluate whether they have experienced a VTE or bleed. For this study no additional hospital visits are necessary.

DETAILED DESCRIPTION:
Background

Total hip arthroplasty (THA) and total knee arthroplasty (TKA) are associated with an overall symptomatic venous thromboembolism (VTE) risk of about 1.3% despite the use of prophylactic anticoagulants in all patients. While not preventing all VTEs, the uniform application of anticoagulant prophylaxis is at the same time associated with a major bleeding risk of at least 0.5%. Considering that a large proportion of all patients actually have a low VTE risk, this group is unnecessarily exposed to the burden and risks of thrombosis prophylaxis. On the contrary, some patients with a high VTE risk experience a VTE despite the use of the same prophylactic anticoagulants. These VTE cases could have possibly been prevented by intensified prophylaxis.

Objectives

Overall objective: To study whether the application of a targeted anticoagulation strategy leads to less thrombotic and bleeding complications in this large patient group.

Primary objective DISTINCT study arm 1 : To determine whether in-hospital thrombosis prophylaxis only is as effective compared with the standard thrombosis prophylaxis approach to prevent symptomatic VTE after total knee and hip arthroplasty in patients with a low VTE risk.

Primary objective DISTINCT study arm 2: To determine the incidence of symptomatic VTE after total knee and hip arthroplasty in patients with an intermediate VTE risk.

Primary objective DISTINCT study arm 3: To determine whether intensified thrombosis prophylaxis is more effective and equally safe compared with standard thrombosis prophylaxis to prevent symptomatic VTE in patients with a high VTE risk by comparing symptomatic VTE and bleeding complications.

Methods

The investigators hypothesize that:

1. In patients with a low VTE risk the thromboprophylaxis can be safely shortened to in-hospital duration only, without increasing the VTE risk (in comparison with the standard duration). In addition, this will lead to less bleeds.
2. In patients with a high VTE risk (individual predicted risk >1.5%), a therapeutic dose of thrombosis prophylaxis for 6 weeks is more effective to prevent symptomatic VTE, in comparison with the standard thromboprophylaxis. In addition, the investigators expect that the benefits of this approach (less symptomatic VTEs) outweigh the induced bleeds.

In the trial participants are allocated to one of three study arms based on the postoperative venous thromboembolism (VTE) risk predicted with the TRiP(plasty) score. (Nemeth, 2024)

* DISTINCT 1 (low VTE risk, <1.0%) will be a randomized study arm.
* DISTINCT 2 (intermediate VTE risk, 1.0%-1.5%) will be an observational study arm.
* DISTINCT 3 (high VTE risk, >1.5%) will be a randomized study arm.

Participants will receive a questionnaire before surgery and 2 weeks, 6 weeks and 3 months after surgery. To assess the outcome measures. Furthermore an additional questionnaire is send 1 year after surgery if the participant experienced a VTE, major bleed or prosthesis infection. This questionnaire is focused on quality of life and joint function. Participants without such an event can be invited to complete this questionnaire as well. No extra hospital visits are needed and the surgery does not change.

Sample size calculations

In DISTINCT study arm 1, the expected 3-month cumulative incidence of symptomatic VTE in the control arm is 0.75%. No risk reduction or increase is anticipated, so the expected risk in the short-duration prophylaxis group is also 0.75%. With a non-inferiority limit set at 1%, a sample size of 3,130 patients is needed to achieve a power of 90%, leading to an aim to include 1,739 patients in each group, totaling 3,478 patients after accounting for a maximum dropout rate of 10%.

For DISTINCT study arm 2, in the intermediate-risk group, the expected cumulative incidence of VTE within 3 months is 1.3%. With a sample size of 2,500, a 95% confidence interval width of 0.9% - 1.7% is expected, ensuring a probability of less than 15% that the upper bound of a two-sided 95% confidence interval will exceed the 2% margin.

In DISTINCT study arm 3, a 3-month cumulative incidence of symptomatic VTE of 2.5% is expected in the control group. With an anticipated relative risk reduction of 50% in the intervention group, a sample size of 3,694 patients is necessary to achieve 80% power. Considering an interim analysis and a slightly stricter statistical significance level at the final analysis, a total of 3,748 patients is required, with 2,050 patients in each arm after accounting for a maximum dropout rate of approximately 9%, totalling 4,100 patients.

Ethics: The study has been approved by the Medical Ethics Committee Leiden Den Haag Delft. All participants will provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo an elective total hip arthroplasty or total knee arthroplasty
* Aged 18 years or older

Exclusion Criteria:

* Primary arthroplasty for fractures
* Revision surgery
* Hemiarthroplasty
* Pregnancy
* Current use of therapeutic anticoagulant therapy of any type (e.g., LMWH, DOAC, vitamin K antagonist)
* A contraindication for either study drug
* Insufficient knowledge of the Dutch language
* Insufficient mental or physical ability to fulfil trial requirements
* Active malignancy (i.e. cancer diagnosis within six months before surgery (excluding basal-cell or squamous-cell carcinoma of the skin), recently recurrent or progressive cancer or any cancer that required anti-cancer treatment within six months before surgery)
* Patients using thrombocyte aggregation inhibitors that cannot be temporarily discontinued at the discretion of their treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10078 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolic events | 90 days postoperative
  Number of VTEs in the first 3 months postoperative.
Major bleeding | 90 days postoperative
  Number of major bleeds in the first 3 months postoperative.

SECONDARY OUTCOMES:
Clinically relevant non major bleeding | 90 days postoperative
  Incidence of clinically relevant non-major bleeding
Impact of events on QALY's | 90 days and 1 year postoperative
  Estimated using the EQ-5D-5L
Healthcare costs | 90 days and 1 year postoperative
  Healthcare costs will be estimated from patient questionnaires at 0, 2, 6, 13 and 52 weeks.
Prosthetic joint infections | 90 days postoperative
  Defined according to the European Bone and Joint Infection Society (EBJIS) definition of periprosthetic joint infection described in Bone Joint J 2021;103-B(1):18-25.
Patient reported quality of life | 90 days and 1 year postoperative
  Measured using the EQ-5D-5L (scored as described in: Value in Health 2016, 19(4), 343-352.)
Patient reported quality of life | 1 year postoperative
  Measured using the 36-Item Short Form Health Survey (score 0-100 with a higher score indicating a higher quality of life)
Patient reported outcome measures | 1 year postoperative
  Measured using Oxford Hip score or Ofxord Knee Score depending on the performed surgery. (score 0-100 with a higher score indicating a better outcome)
Myocardial infarction | 90 days postoperative
  Incidence of myocardial infarction
Ischemic stroke | 90 days postoperative
  Incidence of ischemic stroke
Death | 90 days postoperative
  Incidence of death

CONTACTS AND LOCATIONS:
Overall Officials: Banne Nemeth, dr, Principal Investigator — Leiden University Medical Center
Locations (10):
- Netherlands (10):
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Zuyderland, Geleen, Limburg
  - Anna Ziekenhuis, Geldrop, North Brabant
  - Bravis ziekenhuis, Roosendaal, North Brabant
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg, North Brabant
  - OLVG, Amsterdam, North Holland
  - Bergman Clinics, Naarden, North Holland
  - Isala ziekenhuis, Zwolle, Overijssel
  - Alrijne, Leiderdorp, South Holland
  - Reinier Haga Orthopedisch Centrum, Zoetermeer, South Holland

IPD SHARING:
Plan to Share IPD: Yes
After data collection and data cleaning are finished deidentified data will be registered in a repository and be made available for further research upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Nemeth B, Smeets M, Pedersen AB, Kristiansen EB, Nelissen R, Whyte M, Roberts L, de Lusignan S, le Cessie S, Cannegieter S, Arya R. Development and validation of a clinical prediction model for 90-day venous thromboembolism risk following total hip and total knee arthroplasty: a multinational study. J Thromb Haemost. 2024 Jan;22(1):238-248. doi: 10.1016/j.jtha.2023.09.033. Epub 2023 Nov 22. PMID 38030547
- [Derived] Kok RY, van Bodegom-Vos L, Ettema HB, Groenwold RHH, van den Hout WB, Huisman MV, Klok FA, Nelissen RGHH, van Rein N, van Veen M, Vehmeijer SBW, Wiegerinck JJI, Cannegieter SC, Nemeth B. Study protocol for the DISTINCT trial: inDividual, targeted thrombosIS prophylaxis versus the standard 'one-size-fits-all' approach in patients undergoing Total hIp or total kNee replaCemenT - a national, multicentre, randomised, multiarm, open-label trial. BMJ Open. 2025 Oct 6;15(10):e101180. doi: 10.1136/bmjopen-2025-101180. PMID 41057196